CLINICAL TRIAL: NCT02165657
Title: Effects of UVB Excimer Laser on Serum Inflammatory Markers in Patients With Psoriasis
Brief Title: Excimer Laser, Serum Markers & Psoriasis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants into trial
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Photomedex (Unknown)
Responsible Party: Principal Investigator, Margaret Bobonich, NP, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-13-33; 06-13-33 (Other: Institutional Review Board (IRB) Number)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis
Keywords: Excimer laser; UVB; Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Excimer laser (Experimental): Excimer laser treatment
  Interventions: Device: Excimer laser treatment

INTERVENTIONS:
Device: Excimer laser treatment — Excimer laser irradiation twice a week for up to 20 treatments.

SUMMARY:
The overall aims for this study are to determine whether UVB excimer laser treatment of psoriasis affects serum inflammatory markers, and to assess hyperpigmentation and erythema with excimer laser treatment.

The investigators hypothesize that treatment of psoriasis with UVB delivered via 308 nm excimer laser will decrease the levels of serum inflammatory markers. The investigators hypothesize that treatment will decrease plaque erythema and will result in minimal hyperpigmentation.

DETAILED DESCRIPTION:
Subjects will undergo Excimer treatment twice a week until they reach a PASI 75 improvement, or until they reach the maximum of 20 total treatments. A blood draw to assess serum inflammatory markers will be performed at the screening visit and final visit. Chromameter assessment, photographs, PASI and PGA (Physician Global Assessment) will be performed throughout the study to monitor psoriasis improvement, hyperpigmentation and erythema.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Male or female with diagnosis of psoriasis
* Psoriasis involvement of 5-15% BSA
* Has been off systemic psoriasis therapies (e.g. retinoids, methotrexate, biologic agents, etc) for at least 4 weeks
* Has been off topical therapies (e.g. calcipotriene, topical steroids) for at least 2 weeks
* Fitzpatrick Skin Types I-VI

Exclusion Criteria:

* Active history of photosensitivity (e.g. xeroderma pigmentosum, lupus erythematosus, porphyria, severe polymorphous light eruption, solar urticaria)
* Any suspicion that the psoriasis is of the photosensitive variant.
* Any medical condition that could be aggravated or may cause extreme discomfort during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in serum inflammatory markers | 23 visits (~12 weeks)
  Change in CRP, MPO, S100 and Resistin levels from screening to final visit.

SECONDARY OUTCOMES:
Objective measure of hyperpigmentation | 23 visits (~12 weeks)
  Chromameter Assessment to measure hyperpigmentation. L* values are measured with a chromameter. A lower L* means more hyperpigmentation.
Objective measure of erythema | 23 visits (~12 weeks)
  Chromameter Assessment to measure erythema. a* values are measured with a chromameter. A higher a* means more erythema.
Improvement in Psoriasis based on PASI assessment | 23 visits (~12 weeks)
  PASI will be performed throughout the study to assess response to treatment.
Improvement in psoriasis based on PGA | 23 visits (~12 weeks)
  PGA (Physician Global Assessment) will be performed throughout the study to assess response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Bobonich, NP, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center (Concord Site), Concord, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02165657/Prot_SAP_000.pdf